CLINICAL TRIAL: NCT01172275
Title: Double-Blind, Placebo-Controlled Trial of N-acetylcysteine (NAC) for the Treatment of Pediatric Obsessive-Compulsive Disorder
Brief Title: N-acetylcysteine (NAC) for Pediatric Obsessive-Compulsive Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1004006623
Record Dates: First submitted 2010-07-27; First posted 2010-07-29 (Estimated); Results first posted 2019-09-06 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-08

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Obsessive-Compulsive Disorder; OCD
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- N-Acetylcysteine (Experimental): N-Acetylcysteine effervescent tablets. 1 900mg tablet once a day for 1 week, then 1 900mg tablet twice a day for 1 week and then 1 900mg tablet three times a day for the remaining 10 weeks of the trial.
  Interventions: Drug: N-Acetylcysteine
- Placebo (Placebo Comparator): Placebo effervescent tablets. 1 900mg tablet once a day for 1 week, then 1 900mg tablet twice a day for 1 week and then 1 900mg tablet three times a day for the remaining 10 weeks of the trial. Children receiving placebo will be offered the active intervention after the double-blind portion of the trial.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: N-Acetylcysteine — 1 900mg tablet once a day for 1 week, then 1 900mg tablet twice a day for 1 week and then 1 900mg tablet three times a day for the remaining 10 weeks of the trial.
  Other Names: PharmaNAC
  Arms: N-Acetylcysteine
Other: Placebo — 1 900mg tablet once a day for 1 week, then 1 900mg tablet twice a day for 1 week and then 1 900mg tablet three times a day for the remaining 10 weeks of the trial. Children receiving placebo will be offered the active intervention after the double-blind portion of the trial.
  Arms: Placebo

SUMMARY:
Pediatric Obsessive-Compulsive Disorder (OCD) affects 1-3% of children. The investigators currently have effective first-line interventions for pediatric OCD such as Cognitive Behavioral Therapy (CBT) and pharmacotherapy with serotonin reuptake inhibitors (SRIs). However, roughly half of children with OCD still have clinically significant OCD symptoms despite treatment with first-line pharmacological treatments and CBT interventions for OCD. Furthermore, all pharmacological treatments for OCD in children have an increased side effect burden when compared to adults. Novel treatments for children with OCD are needed.

N-acetylcysteine (NAC) is a natural supplement that acts as an antioxidant and a glutamate modulating agent. NAC has been used safely for decades in doses 20-40 times higher than in this trial as an antidote for acetaminophen overdose. The only side-effect commonly seen with NAC is nausea and this side-effect is seldom seen in the doses used in this trial.

NAC has recently been demonstrated to be effective in a double-blind, placebo-controlled trial in adults with trichotillomania (chronic hair pulling). Trichotillomania is an obsessive-compulsive spectrum disorder that is hypothesized to be closely related to OCD. In other trials NAC has evidence of some efficacy in treating diverse psychiatric conditions such as bipolar depression, schizophrenia and cocaine dependence.

The investigators are conducting this trial to determine if NAC is effective in treating OCD.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 8-17 years.
* Primary diagnosis of OCD.
* Duration of OCD greater than 6 months.
* Significant Current OCD symptoms: Current CY-BOCS score > or = 16.

Exclusion Criteria:

* Comorbid bipolar disorder, psychotic disorder, substance use disorder, developmental disorder or mental retardation (IQ<70).
* Recent change (less than 4 weeks) in medications that have potential effects on OCD severity (such as Selective Serotonin Reuptake Inhibitors, clomipramine, naltrexone, lithium, psychostimulants, anxiolytics, or antipsychotics). Medication change is defined to include either dose changes or medication discontinuation.
* Recent change in behavioral treatment for OCD or comorbid conditions within the last 4 weeks or initiation of behavioral therapy for tics within the last 12 weeks.
* Asthma requiring medication use within the last 3 months (case reports have linked intravenous NAC administration with asthma exacerbation)
* Known hypersensitivity or previous anaphylactoid reaction to acetylcysteine or any components in its preparation.
* Positive pregnancy test or drug screening test.
* Previous use of N-acetylcysteine (dose greater than 600mg for more than 2 weeks).
* Previous history or suspicion of cystinuria because of a possibility of forming kidney stones.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 11 (Actual)
Dates: Start 2012-07; Primary Completion 2017-02-13 (Actual); Study Completion 2018-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael H. Bloch, MD, MS, Principal Investigator — Yale University
Locations (1):
- Yale Child Study Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lafleur DL, Pittenger C, Kelmendi B, Gardner T, Wasylink S, Malison RT, Sanacora G, Krystal JH, Coric V. N-acetylcysteine augmentation in serotonin reuptake inhibitor refractory obsessive-compulsive disorder. Psychopharmacology (Berl). 2006 Jan;184(2):254-6. doi: 10.1007/s00213-005-0246-6. Epub 2005 Dec 22. PMID 16374600
- [Background] Grant JE, Odlaug BL, Kim SW. N-acetylcysteine, a glutamate modulator, in the treatment of trichotillomania: a double-blind, placebo-controlled study. Arch Gen Psychiatry. 2009 Jul;66(7):756-63. doi: 10.1001/archgenpsychiatry.2009.60. PMID 19581567
- [Background] Berk M, Copolov DL, Dean O, Lu K, Jeavons S, Schapkaitz I, Anderson-Hunt M, Bush AI. N-acetyl cysteine for depressive symptoms in bipolar disorder--a double-blind randomized placebo-controlled trial. Biol Psychiatry. 2008 Sep 15;64(6):468-75. doi: 10.1016/j.biopsych.2008.04.022. Epub 2008 Jun 5. PMID 18534556
- [Background] Berk M, Copolov D, Dean O, Lu K, Jeavons S, Schapkaitz I, Anderson-Hunt M, Judd F, Katz F, Katz P, Ording-Jespersen S, Little J, Conus P, Cuenod M, Do KQ, Bush AI. N-acetyl cysteine as a glutathione precursor for schizophrenia--a double-blind, randomized, placebo-controlled trial. Biol Psychiatry. 2008 Sep 1;64(5):361-8. doi: 10.1016/j.biopsych.2008.03.004. Epub 2008 Apr 23. PMID 18436195
- [Background] Ng F, Berk M, Dean O, Bush AI. Oxidative stress in psychiatric disorders: evidence base and therapeutic implications. Int J Neuropsychopharmacol. 2008 Sep;11(6):851-76. doi: 10.1017/S1461145707008401. Epub 2008 Jan 21. PMID 18205981
- See also: Yale Child Study Center TS/OCD Clinic — http://childstudycenter.yale.edu/ocd/index.html
- See also: Yale OCD Adult Research Clinic — http://psychiatry.yale.edu/research/programs/clinical_people/ocd.aspx

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | N-Acetylcysteine | Placebo
Started | 5 | 6
Completed | 3 | 6
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | N-Acetylcysteine | Placebo | Total
Number analyzed (Participants) | 5 | 6 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5 | 6 | 11
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 6 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: OCD Severity at 12 Weeks
Description: Children's Yale-Brown Obsessive-Compulsive Scale (CY-BOCS) (0-7:Subclinical, 8-15: Mild, 16-23: Moderate, 24-31: Severe, 32-40: Extreme)
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | N-Acetylcysteine | Placebo
Number analyzed (Participants) | 5 | 6
points on a scale | 21.4 (4.65) | 21.3 (4.64)

2. Secondary Outcome: Overall Improvement at 12 Weeks
Description: Clinician Global Improvement Scale (CGI) 0=Not assessed 4=Moderately ill
  1. Normal, not at all ill 5=Markedly ill
  2. Borderline mentally ill 6=Severly ill
  3. Mildly ill 7=Very much worse
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | N-Acetylcysteine | Placebo
Number analyzed (Participants) | 5 | 6
score on a scale | 3.2 (1.16) | 3.5 (0.90)

ADVERSE EVENTS:
Time Frame: Adverse events were collected up until 12 weeks.
Arm/Group | N-Acetylcysteine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/6
Other Adverse Events (participants affected / at risk) | 1/5 | 1/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | N-Acetylcysteine (N=5) | Placebo (N=6)
Skin Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-17): https://cdn.clinicaltrials.gov/large-docs/75/NCT01172275/Prot_SAP_000.pdf